CLINICAL TRIAL: NCT02633553
Title: An Open-label, Multi-center, Randomized Phase III Study of Adjuvant Radiotherapy for Stage II/III Thymoma After Complete Resection
Brief Title: Adjuvant Radiotherapy for Stage II/III Thymoma After Complete Resection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Kailiang Wu, professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1508151-4
Record Dates: First submitted 2015-12-15; First posted 2015-12-17 (Estimated); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Thymoma
Keywords: thymoma; adjuvant radiotherapy; complete resection
MeSH Terms: conditions — Thymoma | interventions — Radiotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- radiotherapy group (Experimental): complete resection and adjuvant radiotherapy
  Interventions: Radiation: adjuvant radiotherapy
- observation group (No Intervention): complete resection

INTERVENTIONS:
Radiation: adjuvant radiotherapy — 50Gy/25Fx
  Other Names: RT
  Arms: radiotherapy group

SUMMARY:
This study is designed to investigate whether adjuvant radiotherapy after complete resection has a better survival for stage II or III thymoma.

DETAILED DESCRIPTION:
It is confirmed by many studies that patients of thymoma with complete resection have better prognosis than those with either incomplete resection or without surgery. However,whether patients with stage II or III thymoma could benefit from adjuvant radiotherapy after complete resection remains controversial. The purpose of this study is to investigate whether adjuvant radiotherapy after complete resection can improve survival for stage II or III thymoma.

ELIGIBILITY:
Inclusion Criteria:

18~75 years old; Eastern Cooperative Oncology Group performance status of 0 to 2; Pathologically confirmed masaoka stage II or III thymoma; Have adequate bone marrow, hepatic, and renal function; Patients receive complete resection within 3 months; Written informed consent.

Exclusion Criteria:

Patients with distant metastases; Patients underwent radiotherapy or chemotherapy; Patients who have malignancy history excluding carcinoma in situ of cervix in the previous five years; Active clinical pulmonary infection; Pregnant or nursing.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2018-01-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
DFS (Disease free survival) | 5 years
  from registration to disease progression or death.

SECONDARY OUTCOMES:
OS(overall survival) | 5 years
  from registration to death
Number of Participants with Treatment- Related Adverse Events as Assessed by CTCAE v4.0 | 5 years
  Adverse Events Assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Kailiang Wu, Shanghai, Shanghai Municipality, China